CLINICAL TRIAL: NCT05792189
Title: Evaluation of the Management of Periprosthetic Distal Femur Fractures and Native Knee Distal Femur Fractures, Comparing Open Reduction Internal Fixation With Distal Femur Replacement, a Prospective Cohort Study
Brief Title: Distal Femur Fx: ORIF(Open Reduction and Internal Fixation) vs DFR (Distal Femur Replacement Total Knee Arthroplasty)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202300246
Record Dates: First submitted 2023-02-28; First posted 2023-03-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Distal Femur Fracture
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Intervention Model Description: Prospective, non randomized study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open reduction and internal fixation (ORIF) of distal femur fracture (Active Comparator): Su Type 2 or 3 periprosthetic distal femur fractures about a total knee after undergoing ORIF for a minimum of 2 years
  Interventions: Other: Timed Up and Go Test on subjects with ORIF of distal femur fractures; Other: Koos Jr assesment on subjects with ORIF of distal femur fractures
- Distal femur replacement total knee arthroplasty (DFR) of distal femur fracture (Active Comparator): Su Type 2 or 3 periprosthetic distal femur fractures about a total knee after undergoing DFR for a minimum of 2 years
  Interventions: Other: Timed Up and Go Test on subjects with DFR of distal femur fracture; Other: Koos Jr assesment on subjects with DFR of distal femur fracture

INTERVENTIONS:
Other: Timed Up and Go Test on subjects with ORIF of distal femur fractures — Subjects will perform the Timed Up and Go Test This test is used to assess mobility. Subjects are asked to wear regular footwear and can use their walking device as needed. Subjects begin by sitting in a standard armchair. Next participants are instructed to walk 10 feet to a designated line at a normal pace. Once they reach the line they are to turn and walk back to the chair and sit down. The test starts on the study staff go signal and ends once the subject is fully seated in the chair. Test will be performed at 6 weeks, 3 months, 6 months, 12 months and 24 months post surgical treatment.
  Arms: Open reduction and internal fixation (ORIF) of distal femur fracture
Other: Koos Jr assesment on subjects with ORIF of distal femur fractures — Subjects will complete the KOOS Jr assessment. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales: symptoms, pain, ADLs, sports/recreation, and quality of life. The maximum score a patient can achieve is 100, indicating no knee problems. The minimum score is zero, indicating severe knee problems.
  Arms: Open reduction and internal fixation (ORIF) of distal femur fracture
Other: Timed Up and Go Test on subjects with DFR of distal femur fracture — Subjects will perform the Timed Up and Go Test This test is used to assess mobility. Subjects are asked to wear regular footwear and can use their walking device as needed. Subjects begin by sitting in a standard armchair. Next participants are instructed to walk 10 feet to a designated line at a normal pace. Once they reach the line they are to turn and walk back to the chair and sit down. The test starts on the study staff go signal and ends once the subject is fully seated in the chair. Test will be performed at 6 weeks, 3 months, 6 months, 12 months and 24 months post surgical treatment.
  Arms: Distal femur replacement total knee arthroplasty (DFR) of distal femur fracture
Other: Koos Jr assesment on subjects with DFR of distal femur fracture — Subjects will complete the KOOS Jr assessment. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales: symptoms, pain, ADLs, sports/recreation, and quality of life. The maximum score a patient can achieve is 100, indicating no knee problems. The minimum score is zero, indicating severe knee problems.
  Arms: Distal femur replacement total knee arthroplasty (DFR) of distal femur fracture

SUMMARY:
Supracondylar femur periprosthetic fractures about a total knee arthroplasty (TKA) are a catastrophic and challenging complication of TKA and unfortunately are increasing in incidence. Fixation of these fractures can be challenging due to altered anatomy for the TKA and the presence of the metallic femoral component and have a relatively high complication rate. As a result, some surgeons elect to treat these fractures with a distal femur replacement total knee arthroplasty (DFR). The purpose of this study is to prospectively evaluate periprosthetic femur fractures treated with ORIF or DFR and compare various outcomes measures (Get up and go times, KOOS Jr score)

DETAILED DESCRIPTION:
Supracondylar femur periprosthetic fractures about a total knee arthroplasty (TKA) are a catastrophic and challenging complication of TKA and unfortunately are increasing in incidence. Fixation of these fractures can be challenging due to altered anatomy for the TKA and the presence of the metallic femoral component and have a relatively high complication rate. As a result, some surgeons elect to treat these fractures with a distal femur replacement total knee arthroplasty (DFR). Several small retrospective studies have compared outcomes with mixed results. To the authors' knowledge there are no prospective studies evaluating the outcomes after treatment of periprosthetic distal femur fractures. The purpose of this study is to prospectively evaluate periprosthetic femur fractures treated with ORIF or DFR and compare various outcomes measures (Get up and go times, KOOS Jr score).

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients
* 55 years or older with Su Type II or Su Type III periprosthetic femur fractures or OTA/OA 33C or 338/3 native knee distal femur fracturing requiring surgical intervention and are medically fit to undergo surgical intervention

Exclusion Criteria:

* Patients with an active total knee prosthetic infection
* Patients unable to undergo surgical intervention
* Patient with an open fracture
* Non-English-speaking patients
* Oncologic/pathologic fracture
* Poly-trauma patient (or other associated major orthopaedic injuries)

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Open reduction and internal fixation (ORIF) of distal femur fracture | Up to 2 years
  Subjects will perform the Timed Up and Go Test, This test is used to assess mobility. Subjects are asked to wear regular footwear and can use their walking device as needed. Subjects begin by sitting in a standard armchair. Next participants are instructed to walk 10 feet to a designated line at a normal pace. Once they reach the line they are to turn and walk back to the chair and sit down. The test starts on the study staff go signal and ends once the subject is fully seated in the chair.

SECONDARY OUTCOMES:
Distal femur replacement total knee arthroplasty (DFR) of distal femur fracture | Up to 2 years
  Subjects will complete the KOOS Jr assessment. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-reported outcome measure assessing the patient's opinion about the health, symptoms, and functionality of their knee. It is a 42-item questionnaire, including 5 subscales: symptoms, pain, ADLs, sports/recreation, and quality of life. The maximum score a patient can achieve is 100, indicating no knee problems. The minimum score is zero, indicating severe knee problems.

CONTACTS AND LOCATIONS:
Locations (1):
- UF & Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Sloan M, Premkumar A, Sheth NP. Projected Volume of Primary Total Joint Arthroplasty in the U.S., 2014 to 2030. J Bone Joint Surg Am. 2018 Sep 5;100(17):1455-1460. doi: 10.2106/JBJS.17.01617. PMID 30180053
- [Background] Hart GP, Kneisl JS, Springer BD, Patt JC, Karunakar MA. Open Reduction vs Distal Femoral Replacement Arthroplasty for Comminuted Distal Femur Fractures in the Patients 70 Years and Older. J Arthroplasty. 2017 Jan;32(1):202-206. doi: 10.1016/j.arth.2016.06.006. Epub 2016 Jun 23. PMID 27449717
- [Background] Wadhwa H, Salazar BP, Goodnough LH, Van Rysselberghe NL, DeBaun MR, Wong HN, Gardner MJ, Bishop JA. Distal Femur Replacement Versus Open Reduction and Internal Fixation for Treatment of Periprosthetic Distal Femur Fractures: A Systematic Review and Meta-Analysis. J Orthop Trauma. 2022 Jan 1;36(1):1-6. doi: 10.1097/BOT.0000000000002141. PMID 34001801
- [Background] Darrith B, Bohl DD, Karadsheh MS, Sporer SM, Berger RA, Levine BR. Periprosthetic Fractures of the Distal Femur: Is Open Reduction and Internal Fixation or Distal Femoral Replacement Superior? J Arthroplasty. 2020 May;35(5):1402-1406. doi: 10.1016/j.arth.2019.12.033. Epub 2019 Dec 20. PMID 31924488